CLINICAL TRIAL: NCT01548989
Title: Validation of a New Sexuality Questionnaire: a Tool for Evaluating the Sexuality of Patients With Urinary Incontinence or Pelvic Organ Prolapse
Brief Title: Validation of a New Sexuality Questionnaire for Patients With Urinary Incontinence or Pelvic Organ Prolapse
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2011/BF-02; 2012-A00134-39 (Other: RCB number)
Record Dates: First submitted 2012-02-29; First posted 2012-03-08 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Pelvic Organ Prolapse; Urinary Incontinence; Fecal Incontinence
Keywords: linguistic validation of a new questionnaire
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence; Fecal Incontinence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The study population: Patients suffering from pelvic organ prolapse and/or urinary incontinence and/or fecal incontinence. See inclusion/exclusion criteria.

SUMMARY:
The main objective of this study is to perform the linguistic validation of a new french questionnaire in a population of sexually active (or not) patients who have undergone surgery (or not) for stress urinary incontinence or genital prolapse.

ELIGIBILITY:
Inclusion Criteria:

* The patient is able to read and understand French
* The patient must be insured or beneficiary of a health insurance plan
* Patients suffering from pelvic organ prolapse and/or urinary incontinence and/or fecal incontinence.

Exclusion Criteria:

* Patient is pregnant
* The patient is under judicial protection, under tutorship or curatorship
* The patient does not understand French

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from pelvic organ prolapse and/or urinary incontinence and/or fecal incontinence.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Patient comprehension | Baseline (Day 0; transversal study)
  These tests assess patient understanding of the original formulation and patient understanding of the various terms used: a list of proposed rewording suggested by patients is made.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Fatton, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard, France